CLINICAL TRIAL: NCT05934981
Title: Randomized Trial Comparing Low Pressure in Laparoscopic Colorectal Resection With Warm and Humidified Carbon Dioxide Pneumoperitoneum Versus Low Pressure Pneumoperitoneum Alone
Brief Title: Laparoscopic Colorectal Surgery Using Low-pressure Combined With Warm and Humidified Carbon Dioxide Insufflation
Acronym: PAROS3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bordeaux Colorectal Institute Academy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCIA 2022/01
Record Dates: First submitted 2023-05-30; First posted 2023-07-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Surgery; Benign or Malignant Rectal or Colon Tumors
Keywords: colorectal pathology; laparoscopic; low pressure; early postoperative rehabilitation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Pressure and warm and humidified CO2 insufflation (Experimental): Low pressure pneumoperitoneum and use warm and humidified CO2 insufflation
  Interventions: Procedure: Laparoscopic surgery under low pressure and warm and humidified CO2 Insufflation
- Low Pressure (Active Comparator): Low pressure pneumoperitoneum
  Interventions: Procedure: Laparoscopic surgery under low pressure and conventional Insufflation

INTERVENTIONS:
Procedure: Laparoscopic surgery under low pressure and warm and humidified CO2 Insufflation — low pressure pneumoperitoneum (5-8mmHg) and use warm (35°C), humidified (95% relative humidity) CO2 insufflation.
  Arms: Low Pressure and warm and humidified CO2 insufflation
Procedure: Laparoscopic surgery under low pressure and conventional Insufflation — low pressure pneumoperitoneum (5-8mmHg), and use standard room temperature with dry insufflation.
  Arms: Low Pressure

SUMMARY:
To improve post-operative recovery, medical device was developed combining low-pressure pneumoperitoneum and heated and humidified Carbon Dioxide (95˚F & 95% RH) during laparoscopic surgery to reduce the harmful effects of cold/dry insufflation.

A double-blind, prospective, randomized, controlled, monocentric trial is designed in the aim to assess the impact of low-pressure pneumoperitoneum with warm and humidified gaz on post-operative pain at 24 hours without taking opioids. It is compared with low-pressure laparoscopy with cold and dry gaz in patients undergoing colorectal surgeries.

DETAILED DESCRIPTION:
Laparoscopy is the gold standard in colorectal surgery with many benefits in term of morbidity, post-operative pain and analgesic consumption. However, the pneumoperitoneum created for the laparoscopy has several negatives impact and limits (specific pain following abdominal distension, visibility, physiological repercussion).

To improve recovery after colorectal laparoscopic surgery it was realized a first study (PAROS 1) which showed that low-pressure laparoscopic colectomy for benign or malign disease was feasible and safe with shorter length of stay (3 vs. 4 days; p=0.001), and decrease post-operative pain (VAS ≤ 3 à H8: 87% vs. 72% ; p=0.039) with reduction of analgesic consumption (step II analgesics: 73% vs. 88% ; p=0.032 and step 3 analgesics: (10% vs.23% ; p=0.042) (Br J Surg. 2021 Aug 19;108(8):998-1005) Simultaneously, the development of humidification medical device, referring to the administration of heated and humidified CO2 during laparoscopic surgery, aims to reduce the effects of cell drying and evaporative heat loss when the body is exposed to cold CO2. and dry during laparoscopic surgery. The state of the CO2 traditionally used during laparoscopic surgery and the ambient air during open surgery is very different from that of the human body, as it directly extracts heat and humidity from the already fragile patient.

The introduction of heated and humidified CO2 provides an environment that reflects the physiological state of the peritoneum.

Added to the benefits of low pressure, the advantages of surgical humidification seem very positive. During surgery, surgical humidification would reduce the incidence of perioperative hypothermia, improve local tissue oxygenation and local tissue perfusion. After surgery, it would improve core body temperature, reduce local peritoneal inflammation, surgical site infection rate and recovery time. The benefits of a warmed and humidified CO2 also seem very positive in terms of reducing postoperative pain and analgesic consumption. In the long term, it would reduce adhesion formation, tumor burden, metastases, and economic cost.

The aim of the study is to assess the impact of low-pressure pneumoperitoneum with warm and humidified CO2 insufflation on post-operative pain without taking opioids, compared with low-pressure laparoscopy with cold and dry gas insufflation.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal surgery for malignant or benign pathology
* Surgery without stoma
* Patient operable by laparoscopy or robot assisted under low pressure pneumoperitoneum
* Age ≥ 18 years old
* Patient affiliated to a social security system or beneficiary of the same
* Informing the patient and obtaining free, informed, and written consent, signed by the patient and his investigator.

Exclusion Criteria:

* Laparotomy procedure
* Total or Subtotal Colectomy
* Transverse segmental colectomy
* Proctectomy with stoma or Total Coloproctectomy
* Procedure associated with colorectal surgery (except appendectomy or liver biopsy)
* Patient with stoma
* Probable realization of a stoma during the operation
* Crohn's disease, Hemorrhagic Rectocolitis (UC) with VAS > 3
* Diverticulitis or Sigmoiditis with VAS > 3
* Endometriosis with VAS >3
* VAS before surgery> 3
* BMI ≥ 30
* ASA ≥ 3 (except if ASA 3 for non-cardiac and/or vascular diseases)
* History of laparotomy
* Emergency surgery
* Pelvic Sepsis or Preoperative Fistula
* Pregnant woman, likely to be, or breastfeeding
* Persons deprived of their liberty or under measure of judicial protection (curators or guardianship) or unable to give their consent
* Persons undergoing psychiatric treatment without their consent
* Persons admitted to a health or social establishment for purposes other than research
* Inability to undergo medical monitoring of the trial for geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pain at 24 hours after the end of the intervention by VAS ≤ 3 without taking opioids (without step 2 and step 3 analgesics). | At 24 hours after the end of surgery
  Pain is evaluated with the Visual Analogue Scale (VAS, from 0 (no pain) to 10 (hurts worst)

SECONDARY OUTCOMES:
Operating time | During surgery
  Operating time
Conversion rate in normal pressure and laparotomy | During surgery
  Conversion rate in normal pressure (12-15mmHg) and laparotomy
Peri-operative Heart Rate | During surgery
  Evaluation of Heart rate at different times during surgery : "after anesthetic intubation", "15 min after insufflation", and "5 min after exsufflation".
Perioperative arterial blood pressure | During surgery
  Evaluation of arterial pressure at different times during surgery : "after anesthetic intubation", "15 min after insufflation", and "5 min after exsufflation"
Peri-operative temperature variations | During surgery
  Evaluation of ambient theatre temperature and body temperature at different times during surgery : "before incision", "15 min after insufflation",then every hour and the last temperature reading at the end of the surgery.
Rate of c-reactive protein | from day 1 to day 4 after the end of surgery
  c-reactive protein levels in serum over 4 days post-surgery
Time to bowel opening and passage of gas | An average of 3 days after the surgery
  Time to bowel opening and passage of gas
Number of patients with medical and/or surgical morbidity | From the end of surgery until 3 months of follow-up
  To analyse the cumulative morbidity at 30 days after surgery and at 3 months of follow-up according to the Clavien-DINDO classification
Number of patients with R0 resection | During Surgery
  Rate of cumulative surgery R0 resection for oncologic surgery
Length of stay in hospital | From the surgery to the end of the hospitalization (max30 days)
  Length of stay in hospital
Number of patients with pain at 30 days | From the end of the surgery until 30 days of follow-up
  Pain was evaluated with the Visual Analogue Scale (VAS, from 0 (no pain) to 10 (hurts worst)) during hospital stay and until 30 days using a patient subject diary every day and immediately before each use of pain medication
Number of patients taking analgesics until 30 days | From the end of the surgery until 30 days of follow up
  To analyse the rate of analgesics using a patient subject diary
Mean Score of the EQ-5D-5L Quality of Life | From randomization until 3 months after surgery
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The questionnaire is a self-report survey that measures quality of life across 5 domains: : mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
  - The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, numbered from 0 to 100.
  ( 100 means "the best health you can imagine" and 0 means "the worst health you can imagine".)
Evaluation of predictive factors of postoperative pain | From the surgery until 30 days of follow up
  Study the predictive factors of postoperative pain (VAS>3), 24 hours and 30 days after the surgery. (Visual Analogue Scale (VAS), from 0 (no pain) to 10 (hurts worst)).
Evaluation of predictive factors of opioid intake | From the surgery until 30 days of follow up
  To identify predictive factors of opioid intake (second step and/or third step of the Who analgesic ladder),24 hours and 30 days after the surgery.
  Comparison of the clinical and perioperative data from patients who did or did not consume opioids after surgery. The differences in proportions will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Quentin DENOST, Study Director — Bordeaux Colorectal Institute Academy
Locations (2):
- France (2):
  - Clinique TIVOLI DUCOS - Bordeaux Colorectal Institute, Bordeaux
  - HOPITAL NORD APHM - Service de Chirurgie Digestive, Marseille

IPD SHARING:
Plan to Share IPD: No